CLINICAL TRIAL: NCT01754428
Title: A Multi-Center, Outpatient, Surveillance Study of Respiratory Syncytial Virus (RSV) Infection and Respiratory Syncytial Virus-related Hospitalizations Among Subjects < 24 Months of Age With a Medically Attended Respiratory Tract Infection
Brief Title: Surveillance Study of Respiratory Syncytial Virus Infection (RSV) in Subjects < 24 Months of Age
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-218-0111
Record Dates: First submitted 2012-12-07; First posted 2012-12-21 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory; Syncytial; Virus; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal swabs
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect clinical outcome and nasal viral load information.

DETAILED DESCRIPTION:
There is no vaccine available to prevent Respiratory Syncytial Virus disease; however, a humanized monoclonal antibody is approved for the prevention of Respiratory Syncytial Virus infection in pediatric patients at high risk of disease (eg, pre-term infants, congenital heart disease, and chronic lung disease). Beyond this high-risk group, infection is common in otherwise healthy infants and can be severe, leading to hospitalization and while uncommon, death. Each year in the United States, approximately 100,000 Respiratory Syncytial Virus-related hospitalizations occur in low risk infants. Currently, treatment of infants suffering from Respiratory Syncytial Virus disease is limited to supportive care with the goal of maintaining adequate oxygenation and nutrition.

The availability of a novel anti-Respiratory Syncytial Virus therapeutic that reduces the number of hospitalizations related to Respiratory Syncytial Virus infection would fulfill an unmet medical need in the pediatric population. For maximum effect, such a treatment should be administered as early as possible in the course of infection. Accordingly, the opportunities for early intervention with an anti-Respiratory Syncytial Virus therapeutic are in the outpatient setting, prior to hospitalization. However, the incidence of Respiratory Syncytial Virus-related hospitalization, as well as the natural history and viral dynamics of Respiratory Syncytial Virus infection, remain undefined in the outpatient setting. A better understanding of the prevalence of Respiratory Syncytial Virus infection and subsequent hospitalization rates among symptomatic infants as well as the early disease course of Respiratory Syncytial Virus infection will help in the design of clinical trials needed to assess the efficacy of an anti-Respiratory Syncytial Virus therapeutic developed by Gilead Sciences.

ELIGIBILITY:
Inclusion Criteria:

* < 24 months of age
* ≥ 35 weeks gestational age at birth
* Signs of acute Respiratory Tract Infection < 5 days
* Ability to contact parent or legal guardian for follow up

Exclusion Criteria:

* Ongoing Respiratory Tract Infection
* Lung disease
* Heart disease
* Respiratory Syncytial Virus medication in the last 6 months
* Participation in a study with investigational medicinal product in the last 28 days

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Outpatient pediatric clinics, urgent care facilities or emergency departments
Sampling Method: Probability Sample
Enrollment: 2432 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Determine the percentage of medically attended Respiratory Syncytial Virus- positive subjects hospitalized for Respiratory Syncytial Virus related symptoms | Up to seven months

SECONDARY OUTCOMES:
Percentage of Respiratory Syncytial Virus-positive subjects who sought medical attention, as a result of the Respiratory Tract Infection, after Visit 1 | Up to seven months

CONTACTS AND LOCATIONS:
Overall Officials: John DeVincenzo, MD, Principal Investigator — University of Tennessee
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital/University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Colorado Denver/Children's Hospital Colorado, Denver, Colorado
  - Pediatrics & Adolescent Medicine, P.A., Marietta, Georgia
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, The Ohio State University College of Medicine, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Advanced Pediatrics, Vienna, Virginia
  - Seattle Children's Hospital, Seattle, Washington